CLINICAL TRIAL: NCT05035901
Title: Geometric-Based Handwriting Intervention: Development, Feasibility and Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202009039RIND
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Elementary Students With Handwriting Difficulties
Keywords: handwriting, legibility, visual perception, occupational therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- visual-perception motor-coordination integration program (Experimental): Visual-perception motor-coordination integration program (CCVPMCI) is a Chinese characteristic-based VMI-focused program involving the most Chinese-handwriting-related skills training. CCVPMCI mainly emphasizes the training role of visual-motor integration. The idea of CCVPMCI program will involve (1) visual motor integration training affiliated with visual perception and motor coordination as warm-up exercise, (2) more focus on visual spatial perception in connect with unique visual structure of Chinese characters, (3) the trace or component elements of Chinese characters as the interesting practice material and (4) appropriate challenge for learning.
  Interventions: Other: visual-perception motor-coordination integration program

INTERVENTIONS:
Other: visual-perception motor-coordination integration program — Visual-perception motor-coordination integration program (CCVPMCI) is a Chinese characteristic-based VMI-focused program involving the most Chinese-handwriting-related skills training. CCVPMCI mainly emphasizes the training role of visual-motor integration. The idea of CCVPMCI program will involve (1) visual motor integration training affiliated with visual perception and motor coordination as warm-up exercise, (2) more focus on visual spatial perception in connect with unique visual structure of Chinese characters, (3) the trace or component elements of Chinese characters as the interesting practice material and (4) appropriate challenge for learning.

SUMMARY:
This study will focus on (1) developing the Chinese characteristic-based VMI-focused program, namely visual-perception motor-coordination integration program (CCVPMCI) involving the most Chinese-handwriting-related skills training and (2) investigating the effectiveness of the CCVPMCI program on handwriting performance in children with handwriting difficulties in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. poorer handwriting performance than the peers referred from teachers.

Exclusion Criteria:

1. severe neurological or pervasive developmental disorders that might directly impeded writing
2. intellectual disability that might directly impeded writing
3. musculoskeletal, or sensory (hearing, vision) disorders that might directly impeded writing
4. difficulty in reading or expressing

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-03-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The change from baseline Chinese Legibility Scale (CLS) at one month and six months | baseline, one month, six months
  Chinese Legibility Scale is the self-develop assessment tool to investigate a child's handwriting legibility objectively. Children will be asked to copied 10 Chinese characters on paper within 2*2cm squares to complete the copying paper. Meanwhile, the performance time will be recorded when the child start writing the firs stoke until finish the last stroke of the last character. These Chinese characters are selected from three versions of current mandarin textbooks according to each grade and those with high-frequency and around the average stroke counts will be chosen. Then, characters can be classified into five types of structures based on the visual similarity of character, including top-down (vertical), left-right (horizontal), P-shaped, L-shaped and enclosed. Ultimately, there are 20 characters in total for each grade with five types evenly. The scale will be scored by a therapist blind to the experiment to decide children's writing legibility.
The change from baseline Chinese Handwriting Evaluation Form (CHEF) at one month and six months | baseline, one month, six months
  The CHEF is an observational assessment designed to objectively measure the handwriting performance of school-aged children. It is composed of 25 items and divided into five main dimensions, including construction, accuracy, direction of the characters, writing speed and pencil grip. Items are descriptions of common writing problems by scored on 5-point Likert scale according to the frequency of the problem.

SECONDARY OUTCOMES:
The change from baseline Developmental Test of Visual Perception - Third Edition (DTVP-3) at one month and six months | baseline, one month, six months
  The DTVP-3 is commonly used as a standardized and norm-referenced test to assess visual perception skills for children aged 4 through 12 . The testing time will range from approximately 20 to 40 minutes depending on the child's ability. It is composed of 5 subscales: eye-hand coordination (EH), copying (CO), figure-ground (FG), visual closure (VC) and form constancy (FC). The result of the five subtests can be combined to form three composites: motor-enhanced visual perception, motor-reduced visual perception, and general visual perception. The first two subtests involve motor-enhanced visual perception skills and are summed together to represent visual-motor integration abilities. The latter three subtests (FG, VC and FC) are non-motor involved and are summed together to represent motor-reduced visual perception. The combination of motor-enhanced and motor-reduced visual perception could be the general visual perception skills.
The change from baseline Beery-Buktenica Developmental Test of Visual-Motor Integration at one month and six months | baseline, one month, six months
  The Beery-Buktenica Developmental Test of Visual-Motor Integration is a standardized, norm-referenced test to assess visual-motor integration. During the test, the child is required to copy a series of geometric designs, and his/her performance is compared with standard criteria and reference designs.
Pediatric Motivation Questionnaire (PMQ) | through study completion, an average of one month
  The PMQ is an activity-based measurement of motivation and is designed to measure motivation and the experience of receiving specific therapeutic activities . The items of PMQ are modified from existing questionnaires Pediatric Motivation Scale and based on tenets of self-determination theory. The PMQ consists 12 items containing three motivation domain: (1) extrinsic motivation, (2) basic psychological needs, and (3) intrinsic motivation by 5-point Likert scale. The PMQ represents the motivation condition through the intervention from children their own view. In addition, several open-ended questions are added in children's version to reflect perspective of children while receiving the VPMCI program to obtain qualitative information.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Department of Occupational Therapy, Taipei, Taiwan